CLINICAL TRIAL: NCT02658175
Title: ISIS 304801-CS7 The APPROACH Open Label Study Volanesorsen (ISIS 304801) An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients With Familial Chylomicronemia Syndrome (FCS)
Brief Title: The Approach Open Label Study: A Study of Volanesorsen (Formerly IONIS-APOCIIIRx) in Participants With Familial Chylomicronemia Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akcea Therapeutics (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 304801-CS7; 2015-003755-21 (EudraCT Number)
Record Dates: First submitted 2016-01-12; First posted 2016-01-18 (Estimated); Results first posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Familial Chylomicronemia Syndrome; Lipoprotein Lipase Deficiency; Hyperlipoproteinemia Type 1
MeSH Terms: conditions — Familial hyperchylomicronemia syndrome; Hyperlipoproteinemia Type I | interventions — ISIS 304801

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (3):
- Treatment-naïve Group (Experimental): Treatment naïve group included combined group of ISIS 304801-CS7 (CS7-New) study participant and participant on placebo in index studies (ISIS 304801-CS6 [NCT02211209] and ISIS 304801-CS16 [NCT02300233]), were to receive 300 mg of volanesorsen as single SC once weekly for Weeks 1-52 of this study. Participants were allowed dose adjustment/dose reduction based on monitoring rules. Following Week 52 visit, participants had option of participating in expanded access program or continuing treatment with 300 mg of volanesorsen as single SC once-weekly for up to additional 52 weeks (Weeks 53-104) and in France participants, up to additional 104 weeks for total of 156 weeks (Weeks 105 to Week 156) until expanded access program was approved and available in their country. Participants who were not participating in expanded access program were to enter 13-week post-treatment (PT) evaluation period and in France, participants not continuing treatment were to enter 26-week PT follow-up period.
  Interventions: Drug: Volanesorsen
- CS6-Volanesorsen (Experimental): Participants with FCS rolling over from the ISIS 304801-CS6 (NCT02211209) index study after receiving volanesorsen, were to receive 300 mg of volanesorsen as a single SC injection once weekly for Weeks 1-52 of this study. Participants were allowed dose adjustment/dose reduction based on monitoring rules. Following the Week 52 visit, participants had the option of participating in an expanded access program or continuing treatment with 300 mg of volanesorsen as a single SC injection once-weekly for up to an additional 52 weeks (Weeks 53-104) and in France participants, up to an additional 104 weeks for total of 156 weeks of treatment (Weeks 105 to Week 156) of this study until an expanded access program was approved and available in their country. Participants who were not participating in an expanded access program were to enter a 13-week post-treatment evaluation period and in France, participants not continuing treatment were to enter a 26-week post-treatment follow-up period.
  Interventions: Drug: Volanesorsen
- CS16-Volanesorsen (Experimental): Participants with FCS rolling over from the ISIS 304801-CS16 (NCT02300233) index study after receiving volanesorsen, were to receive 300 mg of volanesorsen as a single SC injection once weekly for Weeks 1-52 of this study. Participants were allowed dose adjustment/dose reduction based on monitoring rules. Following the Week 52 visit, participants had the option of participating in an expanded access program or continuing treatment with 300 mg of volanesorsen as a single SC injection once-weekly for up to an additional 52 weeks (Weeks 53-104) and in France participants, up to an additional 104 weeks for total of 156 weeks of treatment (Weeks 105 to Week 156) of this study until an expanded access program was approved and available in their country. Participants who were not participating in an expanded access program were to enter a 13-week post-treatment evaluation period and in France, participants not continuing treatment were to enter a 26-week post-treatment follow-up period.
  Interventions: Drug: Volanesorsen

INTERVENTIONS:
Drug: Volanesorsen — 300 mg volanesorsen administered via SC injection.
  Other Names: IONIS-APOCIIIRx; ISIS 304801

SUMMARY:
An open-label study of volanesorsen (ISIS 304801) administered subcutaneously to participants with FCS.

DETAILED DESCRIPTION:
This is a multi-center, open-label study for FCS participants rolling over from the ISIS 304801-CS6 (NCT02211209) index study, FCS participants rolling over from the ISIS 304801-CS16 (NCT02300233) index study and Treatment-naïve group. All participants were to receive volanesorsen 300 milligrams (mg) once per week for 52 weeks. Participants were allowed dose adjustment/dose reduction based on monitoring rules. Participants had the option of continuing dosing for an additional 52 weeks (France: up to an additional 104 weeks for a total of 156 weeks) until an expanded access program was approved and available in their country. Participants who were not participating in an expanded access program were to enter a 13-week (France: 26-week) post-treatment evaluation period.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent to participate in the study (signed and dated) and any authorization required by law.
* Able and willing to participate in a 65-week study.

Group 1 and 2:

* Satisfactory completion of ISIS 304801-CS6 (NCT02211209) or ISIS 304801-CS16 (NCT02300233) index studies with an acceptable safety profile, per Sponsor and Investigator judgment.

Group 3:

* Participants who did not participate in the CS6 or CS16 index studies and meet additional inclusion criteria of FCS may enroll in the study.
* History of chylomicronemia.
* A diagnosis of FCS (Type 1 Hyperlipoproteinemia.)
* Fasting triglycerides greater than or equal to (≥)750 milligrams per deciliter [mg/dL] (8.4 millimoles per liter [mmol/L]) at Screening.

Exclusion Criteria:

* Unwilling to comply with lifestyle requirements for the duration of the study.

Group 1 and 2:

* Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the participant unsuitable for enrollment, or could interfere with the participant participating in or completing the study.

Group 3:

* Diabetes mellitus if newly diagnosed or if hemoglobin A1c (HbA1c)≥ 9.0%.
* Active pancreatitis within 4 weeks of screening.
* Acute Coronary Syndrome within 6 months of screening.
* Major surgery within 3 months of screening.
* Treatment with Glybera therapy within 2 years of screening.
* Have any other conditions in the opinion of the investigator which could interfere with the participant participating in or completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (8):
  - IONIS Investigative Site, Huntington Beach, California
  - IONIS Investigative Site, San Francisco, California
  - IONIS Investigative Site, Boca Raton, Florida
  - IONIS Investigative Site, Boston, Massachusetts
  - IONIS Investigative Site, Philadelphia, Pennsylvania
  - IONIS Investigative Site, Houston, Texas
  - IONIS Investigative Site, Norfolk, Virginia
  - IONIS Investigative Site, Seattle, Washington
- IONIS Investigative Site, São Paulo, Brazil
- Canada (4):
  - IONIS Investigative Site, Vancouver, British Columbia
  - IONIS Investigative Site, Chicoutimi, Quebec
  - IONIS Investigative Site, Montreal, Quebec
  - IONIS Investigative Site, Québec
- France (3):
  - IONIS Investigative Site, Paris, Cedex 13
  - IONIS Investigative Site, Marseille
  - IONIS Investigative Site, Nantes
- Germany (2):
  - IONIS Investigative Site, Berlin
  - IONIS Investigative Site, Cologne
- IONIS Investigative Site, Safed, Israel
- Italy (3):
  - IONIS Investigative Site, Palermo
  - IONIS Investigative Site, Roma
  - IONIS Investigative Site, Rome
- IONIS Investigative Site, Amsterdam-Zuidoost, Netherlands
- IONIS Investigative Site, Cape Town, South Africa
- Spain (5):
  - IONIS Investigative Site, A Coruña
  - IONIS Investigative Site, Barcelona
  - IONIS Investigative Site, Madrid
  - IONIS Investigative Site, Seville
  - IONIS Investigative Site, Zaragoza
- United Kingdom (3):
  - IONIS Investigative Site, Birmingham
  - IONIS Investigative Site, London
  - IONIS Investigative Site, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 19 study centers in Canada, France, Italy, Netherlands, South Africa, Spain, United Kingdom and the United States from 23 December 2015 to 15 January 2020.
Pre-assignment Details: A total of 68 participants were enrolled into this study.
Groups:
- Treatment-naïve Group: Treatment naïve group included combined group of ISIS 304801-CS7 (CS7-New) study participant and participant on placebo in index studies (ISIS 304801-CS6- Placebo [NCT02211209] and ISIS 304801-CS16-Placebo [NCT02300233]), were to receive 300 milligrams (mg) of volanesorsen as a single subcutaneous (SC) injection once weekly for Weeks 1-52 of this study. Participants were allowed dose adjustment/dose reduction based on monitoring rules. Following the Week 52 visit, participants had the option of participating in an expanded access program or continuing treatment with 300 mg of volanesorsen as a single SC injection once-weekly for up to an additional 52 weeks (Weeks 53-104) and in France participants, up to an additional 104 weeks for total of 156 weeks of treatment (Weeks 105 to Week 156) of this study until an expanded access program was approved and available in their country. Participants who were not participating in an expanded access program were to enter a 13-week post-treatment evaluation period and in France, participants not continuing treatment were to enter a 26-week post-treatment follow-up period.
Period: Treatment Period: Weeks 1 to 52
Arm/Group | Treatment-naïve Group | CS6-Volanesorsen | CS16-Volanesorsen
Started | 51 | 14 | 3
Completed | 36 | 7 | 3
Not Completed | 15 | 7 | 0
Not completed — Investigator Judgment | 1 | 0 | 0
Not completed — Voluntary Withdrawal | 6 | 2 | 0
Not completed — Adverse Event or Serious Adverse Event (SAE) | 8 | 5 | 0
Period: 1st Extended Treatment: Weeks 53 to 104
Arm/Group | Treatment-naïve Group | CS6-Volanesorsen | CS16-Volanesorsen
Started | 36 | 7 | 3
Completed | 15 | 5 | 1
Not Completed | 21 | 2 | 2
Not completed — Investigator Judgment | 1 | 0 | 0
Not completed — Voluntary Withdrawal | 4 | 0 | 1
Not completed — Adverse Event or SAE | 7 | 0 | 0
Not completed — Other | 1 | 0 | 1
Not completed — Transferred to Early Access Programs | 8 | 2 | 0
Period: 2nd Extended Treatment: Weeks 105 to156
Arm/Group | Treatment-naïve Group | CS6-Volanesorsen | CS16-Volanesorsen
Started (Only those participants in France who continued into the 2nd extended treatment period.) | 1 | 0 | 1
Completed | 0 | 0 | 0
Not Completed | 1 | 0 | 1
Not completed — Adverse Event or SAE | 0 | 0 | 1
Not completed — Transferred to Commercial Treatment | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who were enrolled and received at least one dose of study drug and who had an open-label study baseline triglyceride (TG) assessment.
Groups:
- Treatment-naïve Group: Treatment naïve group included combined group of ISIS 304801-CS7 (CS7-New) study participant and participant on placebo in index studies (ISIS 304801-CS6- Placebo [NCT02211209] and ISIS 304801-CS16-Placebo [NCT02300233]), were to receive 300 mg of volanesorsen as a single SC injection once weekly for Weeks 1-52 of this study. Participants were allowed dose adjustment/dose reduction based on monitoring rules. Following the Week 52 visit, participants had the option of participating in an expanded access program or continuing treatment with 300 mg of volanesorsen as a single SC injection once-weekly for up to an additional 52 weeks (Weeks 53-104) and in France participants, up to an additional 104 weeks for total of 156 weeks of treatment (Weeks 105 to Week 156) of this study until an expanded access program was approved and available in their country. Participants who were not participating in an expanded access program were to enter a 13-week post-treatment evaluation period and in France, participants not continuing treatment were to enter a 26-week post-treatment follow-up period.
- Total: Total of all reporting groups
Arm/Group | Treatment-naïve Group | CS6-Volanesorsen | CS16-Volanesorsen | Total
Number analyzed (Participants) | 51 | 14 | 3 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (14) | 48 (14) | 48 (11) | 47 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 7 | 2 | 43
  Male | 17 | 7 | 1 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 49 | 14 | 3 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 39 | 11 | 3 | 53
  Race: Asian | 11 | 3 | 0 | 14
  Race: Other Race | 1 | 0 | 0 | 1
Fasting Triglyceride (TG) [Mean (Standard Deviation); unit: milligrams per decilitre (mg/dL)] | 2341 (1193) | 1523 (946) | 2081 (706) | 2161 (1166)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline in Fasting Triglyceride (TG)
Description: Baseline for treatment-naïve group was defined as the average of open-label Day 1 pre-dose assessment and the last measurement prior to open-label Day 1. Baseline for CS6-volanesorsen and CS16-volanesorsen arm groups was defined as the average of index study Day 1 pre-dose assessment and the last measurement prior index study Day 1. The values at the Month 3 analysis time point were defined as the average of the Week 12 (Day 78) and Week 13 (Day 85) fasting assessments. The Month 6 analysis time point was at the end of Month 6, and the values were defined as the average of the Week 25 (Day 169) and Week 26 (Day 176) fasting assessments. The values at the Month 12 analysis time point were defined as the average of the Week 50 (Day 344) and Week 52 (Day 358) fasting assessments.
Time Frame: Baseline and Months 3, 6, and 12
Population: FAS included all participants who were enrolled and received at least one dose of study drug and who had an open-label study baseline TG assessment. Here, "number analyzed" signifies participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment-naïve Group | CS6-Volanesorsen | CS16-Volanesorsen
Number analyzed (Participants) | 51 | 14 | 3
percent change
  Percent Change at Month 3: number analyzed (Participants) | 47 | 14 | 3
  Percent Change at Month 3 | -59.8 (37.0) | -49.2 (34.8) | -64.9 (9.1)
  Percent Change at Month 6: number analyzed (Participants) | 49 | 13 | 3
  Percent Change at Month 6 | -45.5 (42.9) | -54.8 (23.8) | -43.0 (19.7)
  Percent Change at Month 12: number analyzed (Participants) | 45 | 12 | 3
  Percent Change at Month 12 | -36.3 (44.2) | -35.1 (45.6) | -41.6 (36.3)

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE was considered related to the investigational drug product. A TEAE was defined as any AE starting or getting worse on or after the first dose of the study drug.
Time Frame: From first dose of study drug to end of follow-up period [Up to Week 182]
Population: Safety Set included all participants who were enrolled and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-naïve Group | CS6-Volanesorsen | CS16-Volanesorsen
Number analyzed (Participants) | 51 | 14 | 3
Participants | 51 | 14 | 3

ADVERSE EVENTS:
Time Frame: From first dose of study drug to end of follow-up period [Up to Week 182]
Description: Safety Set included all participants who were enrolled and received at least one dose of study drug.
Arm/Group | Treatment-naïve Group | CS6-Volanesorsen | CS16-Volanesorsen
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/14 | 0/3
Serious Adverse Events (participants affected / at risk) | 13/51 | 2/14 | 2/3
Other Adverse Events (participants affected / at risk) | 51/51 | 14/14 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-naïve Group (N=51) | CS6-Volanesorsen (N=14) | CS16-Volanesorsen (N=3)
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendon calcification (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-naïve Group (N=51) | CS6-Volanesorsen (N=14) | CS16-Volanesorsen (N=3)
Injection site erythema (General disorders) | 36 | 7 | 1
Injection site pain (General disorders) | 21 | 3 | 0
Injection site swelling (General disorders) | 14 | 5 | 0
Injection site pruritus (General disorders) | 11 | 4 | 0
Injection site discolouration (General disorders) | 12 | 1 | 1
Injection site induration (General disorders) | 11 | 2 | 1
Pyrexia (General disorders) | 11 | 2 | 0
Fatigue (General disorders) | 7 | 3 | 0
Chills (General disorders) | 6 | 3 | 0
Asthenia (General disorders) | 3 | 2 | 2
Injection site bruising (General disorders) | 5 | 2 | 0
Injection site haematoma (General disorders) | 5 | 1 | 0
Injection site oedema (General disorders) | 5 | 1 | 0
Injection site haemorrhage (General disorders) | 3 | 1 | 0
Pain (General disorders) | 2 | 2 | 0
Injection site hypoaesthesia (General disorders) | 3 | 0 | 0
Injection site reaction (General disorders) | 3 | 0 | 0
Injection site urticaria (General disorders) | 1 | 2 | 0
Peripheral swelling (General disorders) | 3 | 0 | 0
Injection site dryness (General disorders) | 1 | 1 | 0
Cyst (General disorders) | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Injection site mass (General disorders) | 0 | 1 | 0
Local swelling (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 21 | 4 | 0
Influenza (Infections and infestations) | 8 | 5 | 0
Urinary tract infection (Infections and infestations) | 8 | 3 | 0
Bronchitis (Infections and infestations) | 5 | 2 | 1
Gastroenteritis (Infections and infestations) | 5 | 1 | 0
Ear infection (Infections and infestations) | 4 | 1 | 0
Sinusitis (Infections and infestations) | 4 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 14 | 5 | 3
Nausea (Gastrointestinal disorders) | 11 | 4 | 1
Vomiting (Gastrointestinal disorders) | 9 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 7 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 5 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 4 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 12 | 4 | 0
Dizziness (Nervous system disorders) | 5 | 2 | 0
Paraesthesia (Nervous system disorders) | 3 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 3 | 0 | 0
Sciatica (Nervous system disorders) | 2 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Platelet count decreased (Investigations) | 15 | 2 | 0
Alanine aminotransferase increased (Investigations) | 5 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0 | 0
Haemoglobin decreased (Investigations) | 3 | 1 | 0
Haematocrit decreased (Investigations) | 3 | 0 | 0
Cold agglutinins (Investigations) | 0 | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 4 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 2 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 4 | 1 | 0
Albuminuria (Renal and urinary disorders) | 1 | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 2 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 3 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Testicular cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 3 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Immunisation reaction (Immune system disorders) | 2 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Device failure (Product Issues) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT02658175/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT02658175/SAP_001.pdf